CLINICAL TRIAL: NCT00846105
Title: Two-Center Intervention Study to Evaluate the Impact of Rapid Molecular Screening on Nosocomial Transmission of Methicillin-Resistant Staphylococcus Aureus (MRSA).
Brief Title: Efficacy Study of Rapid Test to Prevent Hospital Transmission of Methicillin-Resistant Staphylococcus Aureus (MRSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Professor Marc J. Struelens, Erasme University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Erasme-ULB-P2008/201
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Methicillin Resistance; Staphylococcus Aureus; Staphylococcal Infection
Keywords: methicillin resistant Staphylococcus aureus; MRSA; cross-infection; staphylococcal infection; infection control
MeSH Terms: conditions — Staphylococcal Infections; Cross Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapid PCR screen (Experimental): Rapid PCR screen test for detection of MRSA carriers upon hospital admission
  Interventions: Other: Rapid MRSA PCR test for screening carriers
- Conventional culture (Active Comparator): Conventional culture screen for detection of MRSA carriers upon hospital admission
  Interventions: Other: Rapid MRSA PCR test for screening carriers

INTERVENTIONS:
Other: Rapid MRSA PCR test for screening carriers — In the rapid test intervention arm, all patients admitted to study wards will be sampled within 24 h after admission. To ensure comparison of like with like, sample taking will include: (1) a swab from the anterior nares for PCR testing according to the test manufacturer's instructions; (2) the swab of anterior nares, and swabs from throat, perineum and of any wounds, bladder catheter or intravenous catheter exit site will be processed by conventional testing.
  Other Names: GeneXpert MRSA, Cepheid.; Real-time PCR assay for MRSA

SUMMARY:
The purpose of this study is to evaluate the efficacy of a novel PCR-based laboratory test for rapid detection of MRSA carriers to prevent transmission of MRSA in the Belgian acute care hospital setting.

DETAILED DESCRIPTION:
Methicillin-resistant Staphylococcus aureus (MRSA) strains have become endemic pathogens in acute and chronic healthcare facilities in Belgium. MRSA infection is causing increased public concern as it carries a significant risk of morbidity, mortality and has been linked to substantial excess healthcare costs.

Efficient control of MRSA transmission within healthcare facilities critically depends on screening for and isolation of MRSA carriers among admitted patients. Active surveillance cultures for MRSA are now part of clinical practice recommendations both in Europe and the USA. Indeed, studies have indicated that up to 70 % of the patient reservoir for MRSA among hospitalized patients can only be detected by active sampling of muco-cutaneous colonization sites. There is an urgent public health need for early and reliable detection of carriers of MRSA among patients admitted to healthcare facilities, to inform patient isolation and decontamination procedures, and thereby more effectively control cross-infection

The general objectives of this intervention study to be conducted in two large Belgian hospitals are to measure the impact of rapid (< 3 h) PCR detection of MRSA carriage upon patient admission on shortening the delay to implement contact isolation precautions for carriers and reducing nosocomial MRSA transmission to patients admitted in the same wards.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted for more than 48h to a ward in which evaluation in the previous baseline period met the following:

  * > 80 % compliance with admission and discharge conventional culture screening, for the pooled admissions to all study wards;
  * > 80 % compliance with additional MRSA contact isolation procedures, based on a sample of 50 patient care contact observations per hospital in all study wards;
  * pooled incidence of nosocomial MRSA acquisition ≥ 1.5 new cases /100 at risk admissions in the study wards.

Exclusion Criteria:

* Patients staying 48h or less in the study wards

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7400 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To determine if a ≥ 50 % reduction of incidence of nosocomial MRSA acquisition can be observed after replacing culture by PCR for universal MRSA screening of patients upon admission to high incidence units in two acute care hospitals | 5-10 months

SECONDARY OUTCOMES:
Median time required for detection of MRSA carriage after admission | 5-10 months
Median time required for starting isolation of MRSA carriers | 5-10 months
Number of patient-days of MRSA carrier stay in non-isolated conditions | 5-10 months
MRSA nosocomial infection rate | 5-10 months
MRSA cross-transmission rate | 5-10 months
Sensitivity and specificity of PCR vs conventional MRSA screening by culture | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Struelens, MD, PhD, Principal Investigator — Erasme University Hospital
Locations (2):
- Belgium (2):
  - Algemeen Ziekenhuis Sint-Jan AV, Bruges
  - ULB Hopital Erasme, Brussels

REFERENCES:
- [Background] Struelens MJ, Denis O. Rapid molecular detection of methicillin-resistant Staphylococcus aureus: a cost-effective tool for infection control in critical care? Crit Care. 2006;10(2):128. doi: 10.1186/cc4855. PMID 16563177
- [Derived] Roisin S, Laurent C, Denis O, Dramaix M, Nonhoff C, Hallin M, Byl B, Struelens MJ. Impact of rapid molecular screening at hospital admission on nosocomial transmission of methicillin-resistant Staphylococcus aureus: cluster randomised trial. PLoS One. 2014 May 16;9(5):e96310. doi: 10.1371/journal.pone.0096310. eCollection 2014. PMID 24836438